CLINICAL TRIAL: NCT02710513
Title: Technological and Clinical Innovative Protocols for the Production of Functional Foods - 6.5 (ProAliFun65)
Brief Title: ProAliFun_6.5_Health Effects of a Functional Pasta Enriched With Barley Beta-glucans on Healthy Subjects
Acronym: ProAliFun65
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliero-Universitaria Consorziale Policlinico di Bari (Other)
Collaborators: University of Bari (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ProAliFun_6.5_CE4372
Record Dates: First submitted 2016-03-07; First posted 2016-03-16 (Estimated); Last update posted 2016-03-17 (Estimated); Status verified 2016-03

CONDITIONS: Healthy
Keywords: beta-glucans; gut microbiota; p-cresyl sulphate (pCS); indoxyl sulphate (IS); short-chain fatty acid (SCFA)
MeSH Terms: interventions — beta-Glucans

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Beta-glucans (Experimental): 2 months run-in period (Mediterranean Diet-based dietary scheme including a daily supply of 100 g of normal pasta) + 2 months intervention period (Mediterranean Diet-based dietary scheme including a daily supply of 100 g of functional pasta providing 3 g of beta-glucans/day)
  Interventions: Dietary Supplement: Beta-glucans

INTERVENTIONS:
Dietary Supplement: Beta-glucans — 2 months Mediterranean Diet-based free diet (run-in) + 2 months Mediterranean Diet-based free diet with a daily supplementation of 100 g of beta-glucans pasta (intervention). Medical visits, dietary counselling with food frequency questionnaires administration, blood, urine and feces collection were performed before (T0) and after (T2) the two months of beta-glucans intervention.
  Other Names: Functional pasta enriched with barley beta-glucans

SUMMARY:
The purpose of this study is to evaluate the healthy properties of a dietary intervention based on an innovative pasta enriched with prebiotic fibers (barley beta-glucans).

The hypothesis is that the gut microbiota and metabolome, the nutritional status, the redox/subclinical inflammation parameters and the markers of cardiovascular risk may improve in healthy subjects.

DETAILED DESCRIPTION:
This clinical trial is a prospective pilot study, lasting 4 months. A target number of 30 healthy individuals meeting inclusion and exclusion criteria, assessed at enrollment, and which have signed the informed consent, will be recruited.

ELIGIBILITY:
Inclusion Criteria:

* healthy subjects
* aged between 30 and 70 years
* BMI between 18.5 and 24.9
* omnivorous diet
* informed consent signed

Exclusion Criteria:

* diabetes type 2
* urine protein > 1g/24h
* antibiotics and probiotics administration by 15 days before the enrollment
* gastrointestinal, celiac, inflammatory systemic and chronic liver diseases
* recent diagnosis of cancer
* corticosteroid or immunosuppressive therapies
* previous major acute cardiovascular pathologies (heart attack, cerebral ictus)
* hyperlipidemia
* consume of alcohol
* psychiatric diseases

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2014-12; Primary Completion 2015-04 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Reduction in non-HDL cholesterol | at the end of the intervention period (2 months)
  Confirmation of beta-glucans properties in reduction of total and LDL cholesterol

SECONDARY OUTCOMES:
Effects on gut microbiota SCFA modulation | at the end of the intervention period (2 months)
  Measurement of fecal levels of short-chain fatty acids (acetate, propionate, butyrate)
Effects on gut microbiota pCS modulation | at the end of the intervention period (2 months)
  Measurement of circulating levels of p-cresyl sulphate
Effects on gut microbiota IS modulation | at the end of the intervention period (2 months)
  Measurement of circulating levels of indoxyl sulphate
Effects on Flow-mediated dilation (FMD) | at the end of the intervention period (2 months)
  Measurement of beta-glucans effect on endothelial function through FMD

CONTACTS AND LOCATIONS:
Overall Officials: Loreto Gesualdo, MD Full Prof, Principal Investigator — Head of the Nephrology, Dialysis and Transplantation Unit "Aldo Moro" University of Bari Azienda Ospedaliero-Universitaria Consorziale "Policlinico"
Locations (1):
- AOUC "Policlinico", Bari, Italy

IPD SHARING:
Plan to Share IPD: Undecided